CLINICAL TRIAL: NCT00200460
Title: A Double-Blind, Multi-Center, Randomized, Placebo-Controlled, Parallel Group Dosing Study Evaluating the Effects of Nebivolol on Blood Pressure in Patients With Mild to Moderate Hypertension
Brief Title: A Study Evaluating the Effects of Nebivolol on Blood Pressure in Hypertensive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Bertek Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEB302
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Hypertension
Keywords: Nebivolol; Hypertension; Beta-Blocker
MeSH Terms: conditions — Hypertension | interventions — Nebivolol

INTERVENTIONS:
Drug: Nebivolol

SUMMARY:
The purpose of this study is to evaluate the effects of various doses of nebivolol in patients with mild to moderate hypertension.

DETAILED DESCRIPTION:
This was a multi-center, randomized, double-blind, parallel group, placebo-controlled study of nebivolol over a range of doses in patients with mild to moderate hypertension. The study consisted of 2 phases: screening/washout/single-blind placebo run-in followed by randomization/double-blind treatment. During the double-blind phase, patients received nebivolol or placebo. Patients had 7 scheduled clinical visits during the study.

ELIGIBILITY:
Inclusion Criteria:

* An average sitting diastolic blood pressure of greater then or equal to 95 mmHg and less then or equal to 109 mmHg at baseline

Exclusion Criteria:

* Recent myocardial infarction or stroke
* Secondary hypertension
* Contraindications to beta-blocker treatment or discontinuation of current antihypertensive therapy
* Pregnancy, nursing, or women of child-bearing potential not using appropriate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 825
Dates: Start 2001-09; Study Completion 2003-03

PRIMARY OUTCOMES:
The change of the average sitting diastolic blood pressure taken at trough drug plasma level at the end of treatment compared to baseline

SECONDARY OUTCOMES:
- Sitting SBP
- Supine SBP and DBP
- Standing SBP and DBP
- Response rate
- Correlation between plasma levels

CONTACTS AND LOCATIONS:
Overall Officials: Betty S. Riggs, MD, MBA, Study Director — Mylan Pharmaceuticals Inc
Locations (1):
- Mylan Pharmaceuticals Inc., Morgantown, West Virginia, United States